CLINICAL TRIAL: NCT06494592
Title: The Exercise and Concussion Health Study (TECHS)
Brief Title: The Exercise and Concussion Health Study
Acronym: TECHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northeastern University (Other)
Responsible Party: Principal Investigator, Timothy Morris, Principal Investigator, Northeastern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-10-15
Record Dates: First submitted 2024-06-25; First posted 2024-07-10 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Concussion, Mild; Concussion, Brain; TBI (Traumatic Brain Injury); TBI
Keywords: Brain; TBI; Concussion
MeSH Terms: conditions — Brain Concussion; Brain Injuries, Traumatic | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise Group (Experimental)
  Interventions: Behavioral: Aerobic Exercise
- Balance Exercise Group (Active Comparator)
  Interventions: Behavioral: Balance Exercise

INTERVENTIONS:
Behavioral: Aerobic Exercise — Participants in the aerobic exercise intervention group will engage in a virtual aerobic exercise intervention three times a week for 12 weeks for a 30-minute session (5 minute warm up, 20 minutes of aerobic exercise, 5 minutes cooldown) and will receive information about the session prior to their appointment. Sessions have a goal of reaching at least 20 minutes of supervised exercise performed at 80% of the heart rate at symptom threshold.
  Arms: Aerobic Exercise Group
Behavioral: Balance Exercise — Participants in the balance exercise intervention group will participate in a staff-led virtual session three times a week for 12 weeks for a 30-minute session and will receive information about the session prior to their appointment. This group will focus on improving balance, with some additional work on flexibility and strength.
  Arms: Balance Exercise Group

SUMMARY:
This study aims to investigate the effect of two different physical exercise interventions on the brain, cognition and patient reported outcomes following a mild traumatic brain injury (mTBI) in community-dwelling adults.

Physical exercise as an intervention for mTBI has great potential yet there is limited high-quality evidence of its effect. Additionally, while standardized exercise protocols for sport-related concussion exist, a similar program is not available to members of the general public who have suffered a mTBI. This study therefore aims to test the effect of a 3-month exercise protocol either focusing on balance or aerobic exercises. The results from the study may lead to advances in evidenced-based mTBI management and provide clinicians with an effective intervention that can improve brain and cognitive recovery after mTBI.

DETAILED DESCRIPTION:
This is a 12-week two arm pilot randomized control trial comparing two types of exercise interventions. Both groups will complete three 30-minute remote exercise sessions weekly, via Zoom delivered by a trained interventionist and supervised by a dedicated safety officer. Participants will be randomly assigned to either aerobic or balance based exercise for the duration of the study. Participants will sign informed consent in person during a baseline visit where measures of brain (magnetic resonance imaging [MRI] and electroencephalography [EEG]), cognition, patient reported outcomes and lifestyle questionnaires are collected. Participants will repeat this session in-person at the end of the 12-week intervention. Participants will wear a wrist-worn Actigraph for 7 consecutive days at 3 time points throughout the intervention period (once each month) to collect daily physical activity levels and sleep metrics. Both interventions will be individualized and progressive in terms of intensity and difficulty. The exercise interventions sessions will be thresholded at a heart rate of 80% symptom threshold assessed at baseline using a modified cycle and fitness test.

ELIGIBILITY:
Inclusion Criteria:

* Suffered from a clinically diagnosed mild traumatic brain injury (concussion) within 1 year of injury.

  *All potential participants who do not have an official concussion diagnosis from a physician or were not recruited directly from Concussion and Brain Injury clinic at Beth Israel Deaconess Medical Center (BIDMC) will have a phone-based consultation with a trained neurologist from BIDMC to confirm a diagnosis of mTBI, (i.e. any loss of consciousness of up to 30 mins, any loss of memory for events immediately before or after the accident for as much as 24h, any alteration in mental state at the time of the accident and a Glasgow coma score of 13 to 15) (Marshall et al., 2012) per a reliance agreement between Beth Israel Deaconess medical center and northeastern university.
* Men and women of all ethnicities/races and socio-economic status.
* 18-55 years.
* Signed Informed consent.
* Physically fit enough to undergo exercise as screened using the Physical Activity Readiness Questionnaire (PAR-Q) and the cardiovascular section of the Health History & Demographics Questionnaire. An affirmative response (i.e., "yes") to any single item regarding an individual's health status is grounds for the necessary medical clearance before enrollment.
* Normal or corrected-to-normal vision based on the minimal 20/20 standard in order to complete the cognitive tasks (below 20/20 vision).
* Able to speak, read, and write English.
* Ambulatory without pain or the assistance of walking devices.
* Reliable means of transportation.
* No diagnosis of a neurological disease.
* MRI compatible.
* No brain bleeds.

Exclusion Criteria:

* Diagnosis of a moderate-to-severe TBI (Glasgow Coma Score of 3-12) or the presentation of skull breach and/or presence of known subdural hematoma.
* Prior diagnosis of cognitive or physical disability (severe asthma, epilepsy, chronic kidney disease, and dependence upon a wheelchair/walking aid).
* Not fluent in English.
* Not medically cleared for exercise.
* Not MRI compatible.
* No history of vasovagal episodes. (sudden drops in heart rate, poor perfusion, constant dizziness)
* History of brain bleeds or strokes.
* Neurological condition (MS, Parkinson's, Dementia, MCI).
* Current treatment for congestive heart failure, angina, uncontrolled arrhythmia, deep-vein thrombosis or other cardiovascular events.
* Myocardial infarction, coronary artery bypass grafting, angioplasty or other cardiac conditions in the past year.
* Regular use of an assisted walking device.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-09-11 (Actual); Study Completion 2025-09-11 (Actual)

PRIMARY OUTCOMES:
Trail Making Test | 12 Weeks
  Cognitive task evaluating executive functioning and processing speed is administered at Baseline and Endpoint at 12 weeks.
Hopkins Verbal Learning Test | 12 Weeks
  Cognitive task evaluating immediate and delayed memory is administered at Baseline and Endpoint at 12 weeks.
Letter and Category Fluency Test | 12 Weeks
  Cognitive task evaluating verbal fluency is administered at Baseline and Endpoint at 12 weeks.

SECONDARY OUTCOMES:
White Matter Diffusion Properties | 12 Weeks
  Completed and analyzed after Baseline and Endpoint via MRI. Diffusion weighted imaging used to measure changes in white matter microstructure.
Resting State Functional Connectivity | 12 Weeks
  Completed and analyzed after Baseline and Endpoint via MRI. Functional MRI scan used to measure changes in resting state brain function via resting state connectivity metrics.
Brain Morphology | 12 Weeks
  Completed and analyzed after Baseline and Endpoint via MRI. Anatomical T1w MRI scan used to measure volume and determine changes in volume over the course of the intervention.
Cerebral Blood Flow | 12 Weeks
  Completed and analyzed after Baseline and Endpoint via MRI. Arterial spin labeling used to measure changes in cerebral blood flow with total cerebral blood flow change.
Electroencephalography (EEG) Power Metrics | 12 Weeks
  From eyes-open and eyes-closed scans: EEG power metrics within the canonical frequency bands (delta, theta, alpha, beta1, beta2, gamma).
EEG Scan- Aperiodic Metrics | 12 Weeks
  From eyes-open and eyes-closed scans: Aperiodic metrics derived from the Fitting Oscillations one over F (FOOOF) algorithm being the aperiodic offset and exponent along with peak power and bandwidth.
Daily Physical Activity Levels- Accelerometers | 12 Weeks
  Wrist-worn Actigraph device is utilized to collect physical activity and sleep metrics at three time points for 7 consecutive days during the 12-week participation.
PROMIS- Patient-Reported Outcomes Measurement Information Systems | 12 Weeks
  Questionnaire collected at Baseline and Endpoint: Self-reported global and cognitive health.
Pittsburgh Sleep Quality Index | 12 Weeks
  Questionnaire collected at Baseline and Endpoint. Self-Reported Questionnaire about sleep duration and quality.
International Physical Activity Questionnaire. | 12 Weeks
  Questionnaire collected at Baseline and Endpoint. Self-reported physical activity measurement.
Symptomology | 12 weeks
  California Interscholastic Federation Graded Concussion Symptom checklist, collected during the baseline session, throughout each intervention session and again at post-test session to assess concussion-related symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Northeastern University, Boston, Massachusetts, United States